CLINICAL TRIAL: NCT02340013
Title: The Effect of Endometrial Shedding With Medroxyprogesterone Acetate Prior to Ovulation Induction With Clomiphene Citrate in Oligo-ovulatory and Anovulatory Women: a Pilot Study
Brief Title: Endometrial Shedding Prior to Ovulation Induction Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-01
Record Dates: First submitted 2014-12-12; First posted 2015-01-16 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medroxyprogesterone acetate (Active Comparator): Medroxyprogesterone acetate 10mg per os x 10 days prior to starting clomiphene citrate 50mg once daily days 3 - 7 of bleeding after stopping medroxyprogesterone acetate
  Interventions: Drug: Medroxyprogesterone acetate
- Control (No Intervention): Women are assigned to start clomiphene citrate 50mg tabs x 5 days on an assigned day, without any vaginal bleeding

INTERVENTIONS:
Drug: Medroxyprogesterone acetate — Women in this arm of the study will be assigned to start medroxyprogesterone acetate 10mg per os x 10 days. This will be followed by vaginal bleeding. On the 3rd day of vaginal bleeding, women will start clomiphene citrate 50mg per os x 5 days for ovulation induction.
  Other Names: Provera
  Arms: Medroxyprogesterone acetate

SUMMARY:
This is a pilot study examining the feasibility of implementing a large randomized control trial looking at the effect of endometrial shedding with medroxyprogesterone acetate compared to no pre-treatment in women taking clomiphene citrate for ovulation induction for infertility due to oligo-ovulation or anovulation.

DETAILED DESCRIPTION:
The purpose of this pilot study is to assess the feasibility of implementing a randomized controlled trial assessing the effect of giving medroxyprogesterone acetate (MPA) to induce a withdrawal bleed compared to a control group of women not receiving MPA on pregnancy rates prior to ovulation induction with clomiphene citrate in oligo-ovulatory and anovulatory women. The primary outcome measure is the effective implementation of the study including a measure of time to recruit 50 patients, physician, nursing and patient compliance rate with the study protocol, and patient satisfaction. Secondary outcome measures include the pregnancy rate per ovulation (where pregnancy is defined as a positive fetal heart rate on ultrasound 2 weeks after a positive pregnancy test), the ovulation rate per cycle started, conception rate per cycle started (where conception is defined as a positive beta-human chorionic gonadotropin level), conception rate per ovulation, time to complete 3 stimulation cycles and endometrial thickness at time of luteinizing hormone surge.

ELIGIBILITY:
Inclusion Criteria:

* Oligo-ovulation defined as having less than or equal to 8 menstrual cycles in the past year or inter-menstrual periods of 45 days or longer
* general good health
* ability to have timed intercourse or intrauterine insemination
* no evidence of tubal dysfunction
* no evidence of a uterine cavity abnormality
* no evidence of male factor infertility

Exclusion Criteria:

* a baseline ultrasound showing an endometrial lining greater than 1.0 cm
* a baseline ultrasound showing an endometrial lining of less than 0.5 cm
* a positive progesterone level at baseline bloodwork
* a positive beta human chorionic gonadotropin level at baseline bloodwork
* body mass index of greater than 40
* women who have previously taken clomiphene citrate for ovulation induction within the last 6 months
* women who are taking metformin
* women who are taking a progestin for luteal phase support.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Composite measure of study feasibility | 2 years
  Time to recruit 50 patients; physician, nursing and patient compliance rate with the study protocol; and patient satisfaction.

SECONDARY OUTCOMES:
pregnancy rate per ovulation | 2 years
ovulation rate per cycle started, | 2 years
conception rate per cycle started | 2 years
conception rate per ovulation | 2 years
time to complete 3 stimulation cycles | 2 years
time to pregnancy | 2 years
endometrial thickness at time of luteinizing hormone surge | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Heather Shapiro, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (2):
- Canada (2):
  - First Steps Fertility, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario